CLINICAL TRIAL: NCT01145807
Title: A Randomized, Double-blind, Vehicle- and Placebo-Controlled, Multicenter Trial in Patients With Mild to Moderate Distal Subungual Toenail Onychomycosis to Investigate the Efficacy, Tolerability, and Safety of Twice Daily Application of TDT 067 for 48 Weeks
Brief Title: TDT 067 Onychomycosis Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Celtic Pharma Development Services (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-067-III-01
Record Dates: First submitted 2010-03-19; First posted 2010-06-17 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Onychomycosis
Keywords: Distal Subungual Toenail Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Terbinafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): non Transfersome® placebo
  Interventions: Drug: Placebo
- Transfersome® vehicle (Sham Comparator): Transfersome® vehicle
  Interventions: Drug: Transfersome
- TDT 067 (Experimental): TDT 067
  Interventions: Drug: TDT067

INTERVENTIONS:
Drug: TDT067 — Study treatment (TDT 067, Transfersome® vehicle, or non Transfersome® placebo) will be applied twice a day for 48 weeks to the great toenail and the other nails and areas surrounding the nails on the foot. Each application will consist of 5 sprays: 1 spray each to the dorsal, medial, anterior, and frontal part of the great toe and a final spray applied evenly to the nail area of the remaining 4 toes. Patients will be instructed not to wash the treated foot or bathe for at least 4 hours after product application.
  Arms: TDT 067
Drug: Placebo — Study treatment (TDT 067, Transfersome® vehicle, or non Transfersome® placebo) will be applied twice a day for 48 weeks to the great toenail and the other nails and areas surrounding the nails on the foot. Each application will consist of 5 sprays: 1 spray each to the dorsal, medial, anterior, and frontal part of the great toe and a final spray applied evenly to the nail area of the remaining 4 toes. Patients will be instructed not to wash the treated foot or bathe for at least 4 hours after product application.
  Arms: Placebo
Drug: Transfersome — Study treatment (TDT 067, Transfersome® vehicle, or non Transfersome® placebo) will be applied twice a day for 48 weeks to the great toenail and the other nails and areas surrounding the nails on the foot. Each application will consist of 5 sprays: 1 spray each to the dorsal, medial, anterior, and frontal part of the great toe and a final spray applied evenly to the nail area of the remaining 4 toes. Patients will be instructed not to wash the treated foot or bathe for at least 4 hours after product application.
  Arms: Transfersome® vehicle

SUMMARY:
The aim of this study is to establish the efficacy, clinical benefits, and safety of treatment with TDT 067 for clinically diagnosed distal subungual onychomycosis of the toenails caused by dermatophytes confirmed by positive mycology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be between 18 and 75 years of age inclusive, of any race, and of either sex.

   Female patients must be either surgically sterile, postmenopausal (no menses for the previous 12 months), or must be practicing an effective method of birth control as determined by the Investigator.
2. Patients must have at least 1 great toenail (target toenail) with clinically diagnosed distal subungual onychomycosis involving between 25% and 65%, inclusive, of the nail and confirmed by KOH visualization and fungal culture positive for dermatophytes. (Patients with culture positive for dermatophytes alone or dermatophytes and non dermatophytes are eligible to participate.) If both great toenails meet inclusion criteria, the one with the greater involvement will be designated the target nail.
3. Patients must be able to understand the requirements of the study, abide by the restrictions, and return for all of the required examinations.
4. Patients must be willing to sign a statement of informed consent.
5. Patients must have a target great toenail with the capability to grow as determined by history of nail cutting.
6. Patients must be willing to refrain from using any nail polish products and other nail cosmetic products on any of the toenails and must be willing to refrain from professional pedicures for the duration of this study.

Exclusion Criteria:

1. Patients who have been treated with an investigational drug within 1 month prior to study start.
2. Patients who are pregnant or planning to become pregnant or who are lactating.
3. Patients with hypersensitivity to terbinafine or to any other ingredients of the formulation.
4. Patients who are unable to spray their toenails and the surrounding tissues on the affected foot without assistance.
5. Patients with symptomatic tinea pedis requiring treatment.
6. Patients using oral terbinafine within 6 months prior to the start of study; patients who have received other oral antifungals within 3 months.
7. Patients using topical antifungal treatments for onychomycosis within 1 month prior to the start of study; patients using topical antifungal treatments for the feet within 1 month prior to the start of the study.
8. Patients with any nail dystrophy that will interfere with the assessment of a clear nail. Patients who have toenail abnormalities or dystrophies that could prevent the restoration of a normal appearing nail in spite of a mycological cure for dermatophytes, including patients with psoriasis, lichen planus, malignancy or pigmentation disorders involving the nail unit, chemical damage, or onychodystrophy due to trauma or other structural deformities.
9. Patients with superficial white or proximal subungual onychomycosis.
10. Patients with a toenail infection involving a non dermatophyte alone.
11. Patients with involvement of the matrix (lunula) or the proximal 2 mm of nail as measured from the proximal nail fold.
12. Patients who have a nail plate with thickness greater than 2 mm or total thickness of the nail plus subungual debris measuring greater than 3 mm.
13. Patients with yellow streaks or dermatophytoma of the target toenail.
14. Patients with a history of peripheral arterial disease or diabetes mellitus.
15. Patients with any condition that in the opinion of the Investigator renders the patient unsuitable for participation in this study.
16. Patients with alanine aminotransferase (ALT) or aspartate (AST) levels greater than 2 times the upper limit of normal without clinical reason, unless, in the opinion of the Investigator, participation in this study would not place the patient at undue risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Cure Rate | 52 Weeks
  To compare complete cure rates for onychomycosis at Week 52 for TDT 067 versus non-Transfersome placebo.
  If the comparison between TDT 067 and non-Transfersome placebo is statistically significant in favor of TDT 067, the following additional primary efficacy objective:
  To compare onychomycosis cure rates at Week 52 for TDT 067 versus Transfersome vehicle

SECONDARY OUTCOMES:
Cure Rate 48 | 48 Weeks
  Compare onychomycosis complete cure rates at Wk 48 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare effective treatment rates at Wk 48 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare mycological cure rates at Wk 48 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare complete cure rates at Wk 48 effective treatment rates at Wks 48, and mycological cure rates at Wks 48 for Transfersome® vehicle versus non Transfersome® placebo
Cure Rate 52 | 52 Weeks
  Compare onychomycosis complete cure rates at Wk 52 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare effective treatment rates at Wk 52 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare mycological cure rates at Wk 52 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare complete cure rates at Wk 52 effective treatment rates at Wk 52 and mycological cure rates at Wk 52 for Transfersome® vehicle versus non Transfersome® placebo
Cure Rate 60 | 60 Weeks
  Compare onychomycosis complete cure rates at Wk 60 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare effective treatment rates at Wk 60 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare mycological cure rates at Wk 60 for TDT 067 versus non Transfersome® placebo and Transfersome® vehicle
  Compare complete cure rates at Wk 60, effective treatment rates at Wk 60, and mycological cure rates at Wk 60 for Transfersome® vehicle versus non Transfersome® placebo

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tschen, MD, Principal Investigator — Academic Dermatology Associates
Locations (1):
- Academic Dermatology Associates, Albequerque, New Mexico, United States